CLINICAL TRIAL: NCT06003530
Title: Phase 1/2a Study for Treatment of Chronic Diabetic Foot Ulcers (DFU) With the Investigational Allogeneic Cell Therapy Product, hOMSC200
Brief Title: Study for Treatment of Chronic Diabetic Foot Ulcers With the Investigational Allogeneic Cell Therapy Product, hOMSC200
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Cytora Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Cyt DFU hOMSC200
Record Dates: First submitted 2023-08-15; First posted 2023-08-22 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Diabetic Foot; Diabetic Foot Ulcer; Diabetic Foot Ulcer Neuropathic
Keywords: diabetic foot ulcer; stem cells
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Intervention Model Description: Patients will be allocated to one of the following arms: Low dose single administration of hOMSC200, High dose single administration of hOMSC200 or Placebo (control) all in addition to SOC treatment
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low dose hOMSC200 (Experimental): Administration of low dose hOMSC200 in addition to routine standard of care
  Interventions: Biological: hOMSC200
- High dose hOMSC200 (Experimental): Administration of high dose hOMSC200 in addition to routine standard of care
  Interventions: Biological: hOMSC200
- Placebo (Placebo Comparator): Administration of placebo in addition to routine standard of care
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: hOMSC200 — Human Oral Mucosal Stem Cells
  Arms: High dose hOMSC200; Low dose hOMSC200
Other: Placebo — Animal component-free, defined cryopreservation medium with 5% DMSO
  Arms: Placebo

SUMMARY:
Purpose of this phase 1/2a study is to assess the safety and efficacy of administration of allogeneic human oral mucosal stem cells (hOMSCs) in patients suffering from chronic diabetic foot ulcers (DFU).

DETAILED DESCRIPTION:
A prospective, placebo controlled, partially blinded and randomized study, comprising two hOMSC200 dose groups (low & high) and one placebo treated group of DFU patients (3 groups; n=8 / treatment groups and n=6/ control group).

Study employs a 2+2 design for dose escalation. The first two patients recruited were treated with a low dose, in a staggered manner, followed by two patients who were recruited to receive the high dose. The remaining patients (18) are randomized to receive the low dose, high dose, or placebo treatment. The assessors and patients will be blinded to the study treatments.

Following administration of hOMSC200 or placebo patients will attend on-site follow up visits for 6 months. During this period safety profile of the investigational product will be assessed as well as measurement of ulcer size. All patients, irrespective of allocated treatment, will receive routine standard of care.

Patients will be followed for long term safety with a phone call interview 1 year following the 6 months termination visit. Optional on-site follow up visits will be offered to all patients during this time period.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Type I or Type 2diabetes and with a neuropathic diabetic foot ulcer for longer than 8 weeks.
* Size of foot ulcer 0.5-13 cm2
* Ulcer graded I by Wager scale
* Ulcer is free of necrotic debris, exhibits no signs of clinical infection
* Ulcer area blood circulation meets one of the following criteria: A. Palpable tibialis anterior and posterior arteries in the affected foot; B. ABI range >0.7 to <1.3; C. TcPO2>30mmHg

Exclusion Criteria:

* Ulcer is of non-diabetic pathophysiology
* The ulcer has decreased in size by >=30% after the screening visit (week -2 to -4 before treatment)
* Severe hepatic deficiency
* Glycated hemoglobin A1C (HbA1C) level of >12%
* Postprandial blood sugar > 350mg/dl
* Require antibiotics to treat the target wound infection within 14 days prior to treatment
* Evidence of current wound infection including pus drainage from wound site
* Severe renal failure (GFR<30) including subject on renal dialysis
* Pregnant or breastfeeding
* Was receiving oral or parenteral corticosteroids, immunosuppressives, or cytotoxic agents prior to 4 weeks from screening
* Patient receiving anticoagulation therapy except for aspirin
* Underwent wound treatments with growth factors, dermal substitutes, or other biological therapies within the last 30 days prior to screening visit

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2022-01-06 (Actual); Primary Completion 2023-12-19 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Treatment related adverse events | 6 months
  Occurrence of treatment-related adverse events assessed by common terminology criteria for adverse events (CTCAE) following recruitment, hOMSC200 administration (ID), and during the follow up.

SECONDARY OUTCOMES:
Wound healing | 24 weeks
  Percentage of wound surface area reduction

CONTACTS AND LOCATIONS:
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel